CLINICAL TRIAL: NCT06152172
Title: CARTIMMUNE: A Single-Center Study of Patients With Autoimmune Diseases Receiving an Autologous Fully-Human Anti-CD19 Chimeric Antigen Receptor T-Cell (KYV 101)
Brief Title: CARTIMMUNE: Study of Patients With Autoimmune Diseases Receiving KYV-101
Acronym: CARTIMMUNE
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: David Porter (Other)
Collaborators: Kyverna Therapeutics (Industry)
Responsible Party: Sponsor-Investigator, David Porter, Director, Cell Therapy and Transplant, University of Pennsylvania, University of Pennsylvania
Organization: University of Pennsylvania (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 855064 - CARTIMMUNE
Record Dates: First submitted 2023-11-21; First posted 2023-11-30 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Idiopathic Inflammatory Myopathies; Diffuse Cutaneous Systemic Sclerosis; SLE Nephritis; ANCA Associated Vasculitis
MeSH Terms: conditions — Myositis; Scleroderma, Diffuse; Lupus Nephritis; Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Intervention Model Description: Participants will be enrolled based on their disease.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- IIM (Experimental): Participants with idiopathic inflammatory myopathy will receive will receive lymphodepleting chemotherapy of cyclophosphamide and fludarabine prior to administration of KYV-101.
  Interventions: Drug: KYV-101; Drug: Cyclophosphamide; Drug: Fludarabine
- DCSS (Experimental): Participants with diffuse cutaneous systemic sclerosis will receive lymphodepleting chemotherapy of cyclophosphamide and fludarabine prior to administration of KYV-101.
  Interventions: Drug: KYV-101; Drug: Cyclophosphamide; Drug: Fludarabine
- SLE (Experimental): Participants with SLE-related nephritis will receive will receive lymphodepleting chemotherapy of cyclophosphamide and fludarabine prior to administration of KYV-101.
  Interventions: Drug: KYV-101; Drug: Cyclophosphamide; Drug: Fludarabine
- AAV (Experimental): Participants with ANCA-associated vasculitis will receive will receive lymphodepleting chemotherapy of cyclophosphamide and fludarabine prior to administration of KYV-101.
  Interventions: Drug: KYV-101; Drug: Cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Drug: KYV-101 — The KYV-101 will be administered IV as a single infusion dosed at 1×108 CAR+ T cells.
Drug: Cyclophosphamide — Lymphodepleting chemotherapy of cyclophosphamide (CYC) 300 mg/m2
Drug: Fludarabine — Lymphodepleting chemotherapy of Fludarabine (FLU) 30 mg/m2 intravenously (IV)

SUMMARY:
The purpose of this study is to assess the safety, tolerability, and clinical activity of KYV 101 (a fully-human anti-CD19 CAR T-cell therapy) in adult subjects with B cell-driven autoimmune diseases. The trial anticipates enrolling participants to reach a maximum of 24 participants who will receive 1 dose of KYV-101 and will be followed for 2 years.

DETAILED DESCRIPTION:
The purpose of this study is to assess the safety, tolerability, and clinical activity of KYV 101 (a fully-human anti-CD19 CAR T-cell therapy) in 24 adult subjects with B cell-driven autoimmune diseases. The diseases under study include: idiopathic necrotizing myopathy (INM) consisting of dermatomyositis (DM), necrotizing myopathy, anti-HMGCoA-associated myopathy, and polymyositis (PM), diffuse cutaneous systemic sclerosis (dcSSc), systemic lupus erythematosus (SLE) with nephritis, and ANCA-associated vasculitis (AAV).

Six participants in each autoimmune disease group for a total of 24 participants will receive a single dose of 1.0×10[8] CAR+ T cells. Participants will be followed under this protocol for 2 years.

Lymphodepleting chemotherapy of cyclophosphamide (CYC) 300 mg/m2 and fludarabine (FLU) 30 mg/m2 intravenously (IV) daily for 3 days will be administered 5 to 7 days prior to administration of KYV-101.

ELIGIBILITY:
Inclusion criteria

Idiopathic inflammatory myopathy (including dermatomyositis, antisynthetase syndrome, immune mediated necrotizing myopathy, and polymyositis):

1. Diagnosis of probable or definite (>55%) idiopathic inflammatory myopathy, including dermatomyositis, anti-synthetase myopathy, immune-mediated necrotizing myopathy (including anti-HMGCoR-myopathy, anti-SRP myopathy), polymyositis, according to the 2017 ACR/EULAR Classification Criteria for idiopathic inflammatory myopathies (Lundberg, Tjarnlund et al. 2017).
2. Disease severity and minimal core set measure criteria: MMT-8 score <136/150, with at least 2 other abnormal core set measures (CSMs) from the following:

   * Patient global VAS≥3 on a 1-10 scale (Appendix 3).
   * Physician's global VAS ≥3 on a 1-10 scale (Appendix 4).
   * Global extramuscular activity score ≥2 cm (Appendix 5).
   * Elevation of at least one of the muscle enzymes (CK, AST, ALT, aldolase, LDH) >1.5 times upper limit of normal (Appendix 6).
   * HAQ-DI ≥0.25 (Appendix 7).
3. Active disease as per one of the following:

   * Creatine kinase ≥4×ULN.
   * Active rashes of dermatomyositis such that CDASI-activity ≥6 (Appendix 8).
   * Evidence on MRI of active myositis within last 6 months.
   * Evidence on EMG of active myositis within last 6 months.
   * Muscle biopsy evidence of active myositis within last 6 months
4. Positive, at screening or by documented medical history, for one myositis-specific per pre specified list (Table 3), except for patients with DM who need not have a positive test for a myositis-specific antibody.

   Table 3. Pre specified List of Autoantibodies

   Myositis-specific: Target Antigen
   * Anti-Jo-1: Histidyl-tRNA synthetase
   * Anti-EJ: Glycyl-tRNA synthetase
   * Anti-PL-7: Threonyl-tRNA synthetase
   * Anti-OJ: Isoleucyl-tRNA synthetase
   * Anti-PL-12: Alanyl-tRNA synthetase
   * Anti-Mi-2: Nucleosome remodeling deacetylase complex
   * Anti-TIF1 gamma; Transcription intermediary factor 1
   * Anti-MDA5: Melanoma differentiation associated protein 5
   * Anti-SAE: Small ubiquitin-like modifier activating enzyme
   * Anti-NXP2: Nuclear matrix protein 2
   * Anti-SRP: Signal recognition particle
   * Anti-HMGCR: 3hydroxy-3methylglutaryl CoA reductase
5. Refractory disease: subject with previous failure (or intolerance) to glucocorticoids and at least two non-glucocorticoids immunosuppressive therapies. An adequate trial of medication defined as at least 12 weeks of therapy or intolerance/adverse reaction necessitating discontinuation.

Diffuse cutaneous systemic sclerosis:

1. Classified as systemic sclerosis according to the 2013 ACR/EULAR classification criteria, with a total score of ≥9.
2. Clinical disease as follows:

   * Classified as diffuse cutaneous SSc.
   * 6 years or less since first non-Raynaud's sign or symptom.
   * Active disease defined as:

     * MRSS ≥16 with, in the prior 6 months, one or more of the following:

       * An increase in MRSS of ≥3 units
       * Involvement of 1 new body area with ≥2 MRSS units
       * 2 new body areas with ≥1 MRSS unit. OR
     * Progressive ILD meeting all of the following criteria

       * Inadequate response or intolerance to at least one treatment, including cyclophosphamide, methotrextate, MMF/mycophenolic acid, nintedanib, rituximab, or tocilizumab.

AND one of the following:

* Evidence of progression on HRCT
* FVC <80%
* DLCO <80%
* evidence of FVC decline of 10% (absolute decline)
* FVC decline of 5% to 9% and DLCO 15%.

SLE-related nephritis:

1. Clinical diagnosis of SLE consistent with the 2019 European League Against Rheumatism (EULAR)/American College of Rheumatology (ACR) classification criteria.
2. Active, biopsy-proven, proliferative LN Class III or IV according to the revised ISN/RPS criteria (Krassanairawiwong, 2021: DOI: 10.1007/s11255-020-02732-3).

   * Overlapping membranous changes are allowed.
   * Biopsy must be within 12 months prior to screening or during screening.
   * Further, the following subjects will be excluded:

     * Significant chronicity defined as: > 50% glomeruli with global sclerosis
     * 50% interstitial fibrosis on renal biopsy
     * 2018 revised International Society of Nephrology (ISN)/Renal Pathology Society (RPS) mNIH chronicity index (CI) ≥5.
3. Inadequate response (Urine Protein ≥1.0 g/24 hours - or equivalent value by spot uPCR but not >7 g/24 hours or equivalent value by spot uPCR) after at least 6 months of treatment with two or more conventional therapies including, but not limited to, belimumab, a calcineurin inhibitor, CYC, mycophenolate mofetil/mycophenolic acid, obinutuzumab, or rituximab.

ANCA-associated vasculitis:

1. Diagnosis of GPA or MPA according to the 2022 ACR/EULAR Classification Criteria.
2. Positive serum PR3-ANCA or MPO-ANCA at screening or by documented medical history.
3. Disease activity/course as follows: Subject must fulfill either A or B

   * A) BVAS/WG ≥3 within prior 60 days (not including the BVAS-WG items of "fever" or "purpura") (Appendix 9) and either:

     * Failure to achieve sustained remission with glucocorticoids and either cyclophosphamide or rituximab given for at least 4 months, OR
     * Intolerance or contraindication to alternative treatments
   * B) Refractory disease defined as:

     * A history of repeated (>2) relapses of AAV despite treatment with immunosuppressive agents OR
     * Requiring prolonged and/or repeated courses of unacceptable doses (as per investigator judgment) of glucocorticoids to maintain adequate control.

Other Inclusion Criteria:

1. Subject must sign a written ICF prior to any screening procedures.
2. Subject must be ≥18 years of age.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2.
4. Adequate organ function as per table below.

Hematology

* Hemoglobin ≥8.5 g/dL without any transfusion support[a]
* Platelets ≥75,000/uL (without transfusion support within 7 days before the laboratory test).
* Absolute Lymphocyte Count (ALC) ≥500/uL (with detectable circulating B cells: >5 cells/mL)
* Absolute Neutrophil Count (ANC) ≥1,200/µL (prior growth factor support is permitted but must be without support in the 7 days prior to the laboratory test)

Hepatic

* AST and ALT ≤2.5×upper limit of normal (ULN)
* Total bilirubin ≤1.5xULN, except in subjects with congenital bilirubinemia, such as Gilbert syndrome (in which case direct bilirubin ≤1.5×ULN is required)

Renal - Creatinine clearance Estimated glomerular filtration rate ≥30 mL/min/1.73 m2 (measured by CKD-EPI Creatinine Equation)

Cardiac

* Left Ventricular Ejection Fraction (LVEF) ≥ 40% confirmed by ECHO/MUGA

  1. For subjects who meet the inclusion criteria at screening, transfusion of red blood cells is permitted after screening as needed to maintain a hemoglobin level ≥8.0 g/dL.

     1. Women of childbearing potential must have a negative pregnancy test at screening using a highly sensitive serum pregnancy test (β-human chorionic gonadotropin [β-hCG]) at screening and prior to lymphodepletion chemotherapy.
     2. Female subjects of childbearing potential who have a fertile male sexual partner must agree to use highly effective methods of contraception (failure rate of <1% per year when used consistently and correctly) specifically 2 forms of contraception, one of which must be a barrier method, from the time of signing the ICF until 1 year after the KYV-101 infusion. Examples of highly effective method of contraception include:

        * Established use of hormonal methods of contraception associated with inhibition of ovulation (eg, oral, inserted, injected, implanted, transdermal), provided the subject or male subject's female partner plans to remain on the same treatment throughout the entire study and has been using that hormonal contraceptive for an adequate period of time to ensure effectiveness.
        * Correctly placed copper containing- intrauterine device or intrauterine hormone-replacing system.
        * Male sterilization with absence of sperm in the post-vasectomy ejaculate.
        * Female sterilization (bilateral tubal ligation/bilateral salpingectomy or bilateral tubal occlusive procedure (provided that occlusion has been confirmed).
        * Sexual abstinence, defined as completely and persistently refraining from all heterosexual intercourse (including during the entire period of risk associated with the study treatments) may obviate the need for contraception ONLY if this is the preferred and usual lifestyle of the subject.
     3. Male subjects, if not surgically sterilized, must agree to use highly effective method of contraception from the time of signing the ICF until 1 year after the KYV-101 infusion.
     4. Women and men must agree not to donate eggs (ova, oocytes) or sperm, respectively, from time of signing the ICF until at least 1 year after receiving a KYV-101 infusion.

     Exclusion Criteria

     Autoimmune Disease-Related Exclusion Criteria

     Idiopathic inflammatory myopathy:

     1a. Evidence of any of the following:
     * Severe muscle damage as per one of the following criteria:

       * Myositis Global Damage Index (MDI) ≥5.
       * Severe proximal muscle atrophy of upper or lower extremity on MRI.
       * Severe proximal muscle atrophy of upper or lower extremity on clinical examination.
       * Wheelchair-bound at home.
       * MMT-8 of ≤80.
     * MDA5-positive rapidly progressing disease (subjects with stable ILD not requiring supplemental oxygen are eligible).
     * Findings of muscular inflammation or myopathy other than the indication, such as inclusion body myositis (IBM), cancer-associated myositis (myositis diagnosed within 2 years of cancer), drug-induced myopathy, amyloid myopathy, muscular dystrophy, metabolic myopathies, or myositis in the context of significant overlap with another systemic autoimmune rheumatologic disease (overlap myositis), except with Sjögren's syndrome.
     * Patients with ILD requiring O2 therapy and/or FVC ≤45% of predicted.
     * Generalized, severe musculoskeletal or neuro-muscular conditions other than IIM that prevent a sufficient assessment of the patient by the physician.

     Diffuse cutaneous systemic sclerosis:

     1.b. Subject with any of the following:

     • Patients with ILD with any of the following
     * Requiring O2 therapy and/or FVC ≤45% of predicted or DLCO ≤40% of predicted at screening
     * Evidence of PAH as defined as estimated RVSP or ≥45 mmHg or right atrial or ventricular enlargement or dilatation, unless subsequent RHC shows no PAH.
     * PAH on right heart catheterization requiring PAH specific treatment.

       • Active bleeding related to gastric antral vascular ectasia (GAVE) in past 6 months.

       • Gastrointestinal dysmotility requiring total parenteral nutrition (TPN).

       • Renal crisis within 1 year prior to enrollment.

       • Pericardial tamponade within 6 months prior to enrollment.

       • Active infection of a digital ulcer within 3 months prior to enrollment.

       • Current gangrene of a digit

     SLE-related nephritis:

     1.c. Subject with any of the following:

     • Evidence of rapidly progressive glomerulonephritis (defined as a doubling of serum creatinine within 3 months prior to enrollment).

     • History of or currently active severe CNS lupus, including cerebritis, cerebrovascular accident (CVA), and seizures. Presence of active neuropsychiatric lupus as assessed by a neurologist and a rheumatologist (at time of screening or during screening period).
     * Patients with volume overload inadequately controlled by a stable dose of diuretics

     ANCA-associated vasculitis:
     1. d. Subject with any of the following acute manifestations of ANCA-associated vasculitis:

        • Alveolar hemorrhage requiring pulmonary ventilation support.

        • Respiratory failure
        * Spinal cord lesion
        * Stroke Abbreviations: CNS=central nervous system; CVA=cerebral vascular accident; DLCO=diffusing capacity of lung for carbon monoxide; FVC=forced vital capacity; ILD=interstitial lung disease; MDI=Myositis Damage Index; MRI=magnetic resonance imaging; PAH=pulmonary arterial hypertension; RHC=right heart catheterization; RSVP=right ventricular systolic pressure

     Other Exclusion Criteria
     1. Prior treatment with cellular immunotherapy (eg, CAR T) or gene therapy product directed at any target.
     2. Positive hepatitis B surface antigen (HBsAg) and hepatitis C serology confirmed by polymerase chain reaction (PCR) (except hepatitis C cured with pharmacotherapy); subjects who are HBsAg negative and hepatitis B core antibody (HBc) positive with no detectable DNA will be allowed into the study but will require regular monitoring of hepatitis B virus (HBV) DNA.
     3. Positive serology for human immunodeficiency virus (HIV).
     4. Primary immunodeficiency.
     5. History of other autoimmune disorders other than the target disease requiring immunosuppressve therapies.
     6. History of stroke, seizure, dementia, Parkinson's disease, coordination movement disorder, cerebellar diseases, psychosis, paresis, aphasia, and any other neurologic disorder investigator considers would increase the risk for the subject.
     7. Subjects who have central nervous system manifestations of the target disease condition i.e., Idiopathic inflammatory myopathy, Diffuse cutaneous systemic sclerosis, SLE, ANCA-associated vasculitis.
     8. Impaired cardiac function or clinically-significant cardiac disease including:

        a. Unstable angina or myocardial infarction or coronary artery bypass graft (CABG) within 6 months prior to leukapheresis.

        b. New York Heart Association (NYHA) stage III or IV congestive heart failure. c. History of clinically significant cardiac arrhythmia (eg, ventricular tachycardia), complete left bundle branch block, high-grade atrioventricular (AV) block.

        d. History of severe ischemic or nonischemic cardiomyopathy. e. Left ventricular ejection fraction (LVEF) <40% as assessed by echocardiogram (ECHO) or multi-gated acquisition (MUGA) scan (performed ≤8 weeks of leukapheresis).
     9. Previous or concurrent malignancy with the following exceptions:

        1. Adequately treated basal cell or squamous cell carcinoma (adequate wound healing is required prior to screening).
        2. In situ carcinoma of the cervix or breast, treated curatively and without evidence of recurrence for at least 3 years prior to screening.
        3. A primary malignancy which has been completely resected, or treated, and is in complete remission for at least 5 years prior to screening.
     10. Serious and/or uncontrolled medical condition that, in the investigator's judgment, would cause unacceptable safety risk, interfere with study procedures or results, or compromise compliance with the protocol, such as:

         1. Active, uncontrolled, viral, bacterial or systemic fungal infection (including human T cell lymphotropic virus [HTLV], human polyomavirus 2 [JC virus], or syphilis); or recent history of repeated infections.
         2. Requirement of supplemental oxygen to maintain oxygen saturation.
         3. Clinical evidence of dementia or altered mental status.
         4. Thromboembolic event within 6 months prior to enrollment
     11. Ongoing toxicity from previous therapy that has not resolved to baseline levels or to Grade 1 or less, except for alopecia, fatigue, nausea, and constipation.
     12. Major surgery planned within 4 weeks prior to leukapheresis or planned within 4 weeks after KYV-101 administration. For surgery planned after 4 weeks post KYV-101 administration, discuss with the sponsor investigator.
     13. Contraindications or life-threatening allergies, hypersensitivity, or intolerance to KYV-101 or its excipients, including dimethyl sulfoxide; or to cyclophosphamide or fludarabine, or to tocilizumab.
     14. Pregnant or breastfeeding; or plans to become pregnant or breastfeed, or father a child within 1 year after receiving the KYV-101 infusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-08-05 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of AEs in IIM. | 3 months after CAR infusion.
  Incidence and severity of AEs in Idiopathic inflammatory myopathies
Incidence and severity of AEs in IIM. | 6 months after CAR infusion.
  Incidence and severity of AEs in Idiopathic inflammatory myopathies.
Incidence and severity of AEs in IIM. | 12 months after CAR infusion.
  Incidence and severity of AEs in Idiopathic inflammatory myopathies.
Incidence and severity of AEs in IIM. | 24 months after CAR infusion.
  Incidence and severity of AEs in Idiopathic inflammatory myopathies.
Incidence and severity of AEs in DCSS | 3 months after CAR infusion.
  Incidence and severity of AEs in diffuse cutaneous systemic sclerosis
Incidence and severity of AEs in DCSS | 6 months after CAR infusion.
  Incidence and severity of AEs in diffuse cutaneous systemic sclerosis
Incidence and severity of AEs in DCSS | 12 months after CAR infusion.
  Incidence and severity of AEs in diffuse cutaneous systemic sclerosis
Incidence and severity of AEs in DCSS | 24 months after CAR infusion.
  Incidence and severity of AEs in diffuse cutaneous systemic sclerosis
Incidence and severity of AEs in SLE Nephritis | 3 months after CAR infusion.
  Incidence and severity of AEs in systemic lupus erythematosus nephritis.
Incidence and severity of AEs in SLE Nephritis | 6 months after CAR infusion.
  Incidence and severity of AEs in systemic lupus erythematosus nephritis.
Incidence and severity of AEs in SLE Nephritis | 12 months after CAR infusion.
  Incidence and severity of AEs in systemic lupus erythematosus nephritis.
Incidence and severity of AEs in SLE Nephritis | 24 months after CAR infusion.
  Incidence and severity of AEs in systemic lupus erythematosus nephritis.
Incidence and severity of AEs in AAV | 3 months after CAR infusion.
  Incidence and severity of AEs in ANCA-Associated vasculitis
Incidence and severity of AEs in AAV | 6 months after CAR infusion.
  Incidence and severity of AEs in ANCA-Associated vasculitis
Incidence and severity of AEs in AAV | 12 months after CAR infusion.
  Incidence and severity of AEs in ANCA-Associated vasculitis
Incidence and severity of AEs in AAV | 24 months after CAR infusion.
  Incidence and severity of AEs in ANCA-Associated vasculitis

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of the Universithy of Pennsylvania, Philadelphia, Pennsylvania, United States